CLINICAL TRIAL: NCT02862990
Title: Evaluation of the Attitude of Pre Menopausal Women With Breast Cancer Faced With the Risk
Brief Title: Evaluation of the Attitude of Pre Menopausal Women With Breast Cancer Faced With the Risk of Fertility Loss Caused by Chemotherapy
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Grupo de Estudios Clínicos Oncológicos Peruano (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0414
Record Dates: First submitted 2016-01-27; First posted 2016-08-11 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Fertility
Keywords: Breast cancer; Fertility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre menopausal women with breast cancer: Pre menopausal women with breast cancer prior treatment in face of infertility evoked by chemotherapy

SUMMARY:
To evaluate the attitude of pre menopausal women with breast cancer faced with the risk of loss of fertility caused by chemotherapy using EORTC's Fertility Questionnaire.

DETAILED DESCRIPTION:
To characterize the attitude of pre menopausal patients with breast cancer regarding the risks of infertility based on the following variables:

* Age at diagnosis
* Number of children
* Will of having children
* Marital status
* Scholarity
* Period of time from the diagnosis
* Time of the last menstruation period
* Chemotherapy administration
* Clinical staging at the diagnosis
* Pathological evaluation
* Documentation of the cancer therapy

ELIGIBILITY:
Inclusion Criteria:

* Women with age ≥ 18 and ≤ 40
* Indication of (neo) adjuvant chemotherapy
* Prior chemotherapy treatment
* Patients with menstrual periods in the last 6 months
* In use of contraceptive methods
* Without breast cancer recurrence
* Capacity to read and understand the informed consent

Exclusion Criteria:

* Patients which received or with indication of definitive ovarian suppression (surgery and/or radiotherapy), except temporary pharmacological ovarian suppression
* Patients whom initiated chemotherapy treatment before entering the study
* Altered state of mind, dementia, or any other psychiatry problem that can interfere in the comprehension or interpretation of the informed consent.
* Previous diagnosis of infertility

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pre menopausal women diagnosed with breast cancer prior treatment
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2015-05; Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
To analyze the number of pre-menopausal patients diagnosed with breast cancer that did not agree in receiving chemotherapy due to the risk of infertility | Baseline and 1 year after after the first interview

SECONDARY OUTCOMES:
Infertility risk for breast cancer patients after accepting chemotherapy | Baseline and 1 year after the first interview
Minimal percentage of cure necessary for patients accept the chemotherapy treatment | Baseline and 1 year after the first interview
Age when diagnosed | Baseline and 1 year after the first interview
Number of children | Baseline and 1 year after the first interview
Desire to have kids | Baseline and 1 year after the first interview
Marital status | Baseline
Scholarity | Baseline
Period of time since the diagnosis | Baseline
Chemotherapy scheme administration | Baseline and 1 year after the first interview
Period of time from the last menstruation period | Baseline and 1 year after the first interview
Description of quality of life of patients with the EORTC QLQ-BR23 | Baseline and 1 year after the first interview

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (7):
- Brazil (3):
  - CPO - Pucrs, Porto Alegre, Rio Grande do Sul
  - HCPA, Porto Alegre, Rio Grande do Sul
  - Hospital Pérola Byington, São Paulo
- Instituto Nacional de Oncologia y Radiobiologia, Havana, Cuba
- Cenro Oncologico Estatal ISSEMYM, Toluca, Mexico
- INEN, Surquillo, Peru
- Hospital de Clínicas San Agustín, Puerto Cabello, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Benson JR, Jatoi I, Keisch M, Esteva FJ, Makris A, Jordan VC. Early breast cancer. Lancet. 2009 Apr 25;373(9673):1463-79. doi: 10.1016/S0140-6736(09)60316-0. PMID 19394537
- [Background] Cardoso F, Loibl S, Pagani O, Graziottin A, Panizza P, Martincich L, Gentilini O, Peccatori F, Fourquet A, Delaloge S, Marotti L, Penault-Llorca F, Kotti-Kitromilidou AM, Rodger A, Harbeck N; European Society of Breast Cancer Specialists. The European Society of Breast Cancer Specialists recommendations for the management of young women with breast cancer. Eur J Cancer. 2012 Dec;48(18):3355-77. doi: 10.1016/j.ejca.2012.10.004. Epub 2012 Oct 29. PMID 23116682
- [Background] Colleoni M, Rotmensz N, Robertson C, Orlando L, Viale G, Renne G, Luini A, Veronesi P, Intra M, Orecchia R, Catalano G, Galimberti V, Nole F, Martinelli G, Goldhirsch A. Very young women (<35 years) with operable breast cancer: features of disease at presentation. Ann Oncol. 2002 Feb;13(2):273-9. doi: 10.1093/annonc/mdf039. PMID 11886005
- [Background] Vallejos Sologuren C, Gómez HL, et al. Clinicopathologic and outcome variables of worse prognosis in premenopausal patients (pts) age 35 and younger. 2010 Breast Cancer Symposium. Abstract 65
- [Background] Reichman BS, Green KB. Breast cancer in young women: effect of chemotherapy on ovarian function, fertility, and birth defects. J Natl Cancer Inst Monogr. 1994;(16):125-9. PMID 7999454
- [Background] Senkus E, Gomez H, Dirix L, Jerusalem G, Murray E, Van Tienhoven G, Westenberg AH, Bottomley A, Rapion J, Bogaerts J, Di Leo A, Neskovic-Konstantinovic Z. Attitudes of young patients with breast cancer toward fertility loss related to adjuvant systemic therapies. EORTC study 10002 BIG 3-98. Psychooncology. 2014 Feb;23(2):173-82. doi: 10.1002/pon.3384. Epub 2013 Aug 29. PMID 24038775
- [Background] Gradishar WJ, Schilsky RL. Ovarian function following radiation and chemotherapy for cancer. Semin Oncol. 1989 Oct;16(5):425-36. No abstract available. PMID 2678491
- [Background] Stearns V, Schneider B, Henry NL, Hayes DF, Flockhart DA. Breast cancer treatment and ovarian failure: risk factors and emerging genetic determinants. Nat Rev Cancer. 2006 Nov;6(11):886-93. doi: 10.1038/nrc1992. Epub 2006 Oct 12. PMID 17036039
- [Background] Dnistrian AM, Schwartz MK, Fracchia AA, Kaufman RJ, Hakes TB, Currie VE. Endocrine consequences of CMF adjuvant therapy in premenopausal and postmenopausal breast cancer patients. Cancer. 1983 Mar 1;51(5):803-7. doi: 10.1002/1097-0142(19830301)51:53.0.co;2-v. PMID 6687378
- [Background] Moore HCF, et al. Phase III trial (Prevention of Early Menopause Study [POEMS]-SWOG S0230) of LHRH analog during chemotherapy (CT) to reduce ovarian failure in earlystage, hormone receptor-negative breast cancer: An international Intergroup trial of SWOG, IBCSG, ECOG, and CALGB (Alliance). J Clin Oncol 32:5s, 2014 (suppl; abstr LBA505)
- [Background] Brandberg Y, Michelson H, Nilsson B, Bolund C, Erikstein B, Hietanen P, Kaasa S, Nilsson J, Wiklund T, Wilking N, Bergh J; Scandinavian Breast Group Study 9401. Quality of life in women with breast cancer during the first year after random assignment to adjuvant treatment with marrow-supported high-dose chemotherapy with cyclophosphamide, thiotepa, and carboplatin or tailored therapy with Fluorouracil, epirubicin, and cyclophosphamide: Scandinavian Breast Group Study 9401. J Clin Oncol. 2003 Oct 1;21(19):3659-64. doi: 10.1200/JCO.2003.07.020. PMID 14512398
- [Derived] Werutsky G, Villarreal-Garza C, Gomez HL, Campos-Gomez S, Reyes RO, Liedke PER, Reinert T, Dybal V, Martinez-Mesa J, Nunes Filho PR, de Jesus RG, Zaffaroni F, Garcia VS, Seibel MF, Barrios P, Rocha MS, Barrios CH. Factors associated with accepting chemotherapy despite the risk of fertility loss in Latin American breast cancer patients-LACOG 0414 study. Ther Adv Med Oncol. 2025 Oct 2;17:17588359251378946. doi: 10.1177/17588359251378946. eCollection 2025. PMID 41049579
- See also: Ferlay J, Shin HR, Bray F, et al. GLOBOCAN 2008 v1.2, Cancer Incidence and Mortality Worldwide: IARC Cancer Base No. 10 [Internet]. Lyon, France: International Agency for Research on Cancer; 2010 — http://globocan.iarc.fr/Default.aspx